CLINICAL TRIAL: NCT04043741
Title: Comparison of Dry Needling and Sustained Pressure in Trigger Points of Lumbar Paraspinal Muscles
Brief Title: Comparison of Dry Needling and Sustained Pressure in Para-spinal Muscles Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Aneela Zia
Record Dates: First submitted 2019-07-30; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Low Back Pain
Keywords: Dry Needling; Oswestry disability index,; Paraspinal muscle length; Pain pressure threshold
MeSH Terms: conditions — Low Back Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant
Masking Description: this study is randomized control trail, participants are randomly allocated through sealed envelope method
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling (Experimental): Dry needling (04 Sessions) and exercises
  Interventions: Other: Dry Needling
- Sustain Pressure (Active Comparator): sustained pressure and Exercises
  Interventions: Other: Sustain Pressure

INTERVENTIONS:
Other: Dry Needling — stretching exercises :single knee to chest (15 reps x 3 sets) double knee to chest(15 reps x 3 sets) strengthening exercises: extension exercises (15 reps x 3 sets)
  Arms: Dry Needling
Other: Sustain Pressure — Sustain Pressure (Number of repetition and hold according to trigger point chronic level)
  + Hot pack 10 to 15 minutes + Active muscle stretching exercise (10 repetition twice daily)
  Arms: Sustain Pressure

SUMMARY:
This study will compare the effect of dry needling and sustained pressure in the lumbar Paraspinal trigger points in terms of pain threshold and muscle length.

There will be two groups ; experimental and control. Half of study group will receive dry needling session along with stretching and strengthening exercises and half of study group will receive sustained pressure technique along with stretching and strengthening exercises .

DETAILED DESCRIPTION:
The study is Randomized Control Trail , which is being conducted in Pakistan Railway hospital and Riphah international hospital (march 2019-june 2019) . Sample size of 50 individual was calculated using epitool with 95% confidence interval (CI), and power 80%. 50 individual are screened out according to inclusion criteria. Individuals are allocated randomly into two groups , 25 in experimental group and 25 in control group by sealed envelope method.Both groups will receive conventional physiotherapy protocol (hot pack, stretching exercises and strengthening exercises) and then experimental group will receive cervical sensorimotor control training. Assessment will be done on baseline, 2nd week, 4th week and 6th week.

Myofascial trigger point (MTrP) is moreover removed or inactivate by means of mechanical stimuli through filiform needle. A swift and repetitious needle insertions into myofascial trigger point is a treatment technique use for dry needling commonly has many therapeutic advantages. It interrupts motor end plates, muscle fibers and distal axons of myofascial trigger points and shortening of related sarcomere of myocytes.

Use of dry needling in combination Muscle Energy Technique (MET) has more significant effects in improving Visual Analog Scale (VAS), Pain Pressure Threshold (PPT) and Range of Motion (ROM) of females patients having latent trigger points in upper trapezius than alone use of MET.

Laser therapy has verified as to be more successful than dry needling in treating MTrPs. It is a preferred option for the patients having apprehensive behavior towards dry needling and health practioners inexpert with the dry needling procedure.

Dry needling is indicated for the treatment when MTrPs are present, may leads to functional restrictions. They are the source of constant peripheral nociceptive contribution which needs to be inactivated. Dry Needling (DN) is also indicated in fascial adhesions, soft tissue restrictions, shortened muscle fiber due to which restricted range of motion is present.Secondary trigger point (TrP) due to different neuromuscular dysfunctions for example in tendonitis, radiculopathies, disk pathology, migraines, carpal tunnel syndrome, tension type headache, joint dysfunction, cranio-mandibular dysfunction, phantom pain , additional regional urological syndromes and other exceptional neurogenic pruritus, Barre Lieou syndrome

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-50.
2. Patient of acute, sub acute, chronic Low back pain (LBP), Mechanical Low back pain (MLBP) and radiculopathies up to one year.
3. Patients having active (spontaneously painful) or latent (requiring palpation to reproduce the characteristic pain) MTrPs.

Exclusion Criteria:

1. Patients that were using any medication to reduce the pain and/or have any effect in the skeletal muscle including analgesics, anticoagulants and muscular relaxants.
2. Taking other treatment in the same period of the research.
3. Pregnant female.
4. Patients with Chronic Disease (kidney disease, Diabetic, and osteoporosis) and spinal diseases (herniated disc, spondylolisthesis) will be excluded.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
The Oswestry Disability Index (ODI) | up to 2 weeks
  Changes from the base line, The Oswestry Disability Index is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools.At the end score is calculated by dividing the obtained score by total (50) multiplied by 100.As one question(section 8) was dropped in all participants ,so total score was considered as 45 instead of 50.
Para-spinal muscle length | up to 2 weeks
  Changes from the base line, Muscle length assessment technique is use to measure available range of muscle. In paraspinal muscles length assessment patient would be sitting position. Palpate anterior superior iliac spine (ASIS) bilaterally and instruct the patient to flex forward producing posterior pelvic tilt. Feel when ASIS starts to move this is the end of thoracolumbar flexion and initiation of posterior pelvic tilt. , Patient forehead would come 10 inches of the knees normally.
Visual analog scale | up to 2 weeks
  Changes from the base line, The visual analogue scale is one dimensional measure of pain intensity in adults inclusive those with chronic pain. The intensity of pain experienced by the patients on this scale range from no pain (score 0) to very severe pain (score 100). It is marked by paper and pencil on a line consist of horizontal (HVAS) or vertical (VVAS) comprised of 10centimeters (100mm) in length.
Pain Pressure Threshold (PPT). | up to 2 weeks
  Changes from the base line, Algometer is a device used to recognize the minimum pressure or force which induce pain pressure threshold (PPT). It is uncomplicated portable tool with a spring install in it. Peak force or pressure provided by this device is kilopond (kp) = 10 N, Newton = 100 kilopascal (kPa).

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Ghafoor Sajjad, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bron C, Dommerholt JD. Etiology of myofascial trigger points. Curr Pain Headache Rep. 2012 Oct;16(5):439-44. doi: 10.1007/s11916-012-0289-4. PMID 22836591
- [Background] Fernandez-de-las-Penas C, Dommerholt J. Myofascial trigger points: peripheral or central phenomenon? Curr Rheumatol Rep. 2014 Jan;16(1):395. doi: 10.1007/s11926-013-0395-2. PMID 24264721
- [Background] Kalichman L, Vulfsons S. Dry needling in the management of musculoskeletal pain. J Am Board Fam Med. 2010 Sep-Oct;23(5):640-6. doi: 10.3122/jabfm.2010.05.090296. PMID 20823359
- [Background] Bishwajit G, Tang S, Yaya S, Feng Z. Participation in physical activity and back pain among an elderly population in South Asia. J Pain Res. 2017 Apr 15;10:905-913. doi: 10.2147/JPR.S133013. eCollection 2017. PMID 28450787
- [Background] Koppenhaver SL, Walker MJ, Su J, McGowen JM, Umlauf L, Harris KD, Ross MD. Changes in lumbar multifidus muscle function and nociceptive sensitivity in low back pain patient responders versus non-responders after dry needling treatment. Man Ther. 2015 Dec;20(6):769-76. doi: 10.1016/j.math.2015.03.003. Epub 2015 Mar 13. PMID 25801100
- [Background] Uemoto L, Nascimento de Azevedo R, Almeida Alfaya T, Nunes Jardim Reis R, Depes de Gouvea CV, Cavalcanti Garcia MA. Myofascial trigger point therapy: laser therapy and dry needling. Curr Pain Headache Rep. 2013 Sep;17(9):357. doi: 10.1007/s11916-013-0357-4. PMID 23904202
- [Background] Desai MJ, Bean MC, Heckman TW, Jayaseelan D, Moats N, Nava A. Treatment of myofascial pain. Pain Manag. 2013 Jan;3(1):67-79. doi: 10.2217/pmt.12.78. PMID 24645933